CLINICAL TRIAL: NCT02338635
Title: Effect of Ursodeoxycholic Acid on Peritoneal Function in Patients on Peritoneal Dialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Duk-Hee Kang, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URSA-1
Record Dates: First submitted 2015-01-12; First posted 2015-01-14 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: End-Stage Kidney Disease
Keywords: ER stress; Peritoneal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- URSA group (Experimental): Drug: Ursodeoxycholic acid Other Name: URSAⓇ (Daewoong Pharmaceutical Co., Ltd) Ursodeoxycholic acid (100 mg/tablet) 300 mg/day ( 100mg tid) for 6 months 3 times after meal
  Interventions: Drug: Ursodeoxycholic Acid
- Placebo group (Placebo Comparator): Placebo drug 1 tablet tid for 6 months

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — Inhibition of ER stress (Ursodeoxycholic Acid)
  Other Names: URSA
  Arms: URSA group

SUMMARY:
Peritoneal fibrosis is one of the major causes of technical failure in patients on peritoneal dialysis (PD) for long period of time. Although the exact mechanisms of peritoneal damage during PD still remain unclear, generation of Endoplasmic reticulum (ER) stress may be responsible for progressive membrane dysfunction. Ursodeoxycholic acid (URSA) is a powerful inhibitor of ER stress to protect peritoneal fibrosis in peritoneal dialysis in the investigators in-vitro study. In this study the researchers investigated the hypothesis that URSA protect peritoneal membrane damage.

DETAILED DESCRIPTION:
Ursodeoxycholic acid (URSA) is known to be relatively safe and beneficial in peritoneal dialysis patient at a dose of 300 mg per day. Patients will be randomly assigned to URSA and placebo group and prescribed according to the protocol. At 2 and 6 month, Peritoneal equilibrium test (PET) will be performed with blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance peritoneal dialysis at least 3 months
* Patients who are able and willing to understand, sign and date an informed consent document, and authorize access to protected health information

Exclusion Criteria:

* Episode of peritonitis at least 3 months
* Episodes of admission due to other disease at lease 3 months
* Liver disease
* Allergic history with Ursodeoxycholic acid
* Nausea or vomiting after Ursodeoxycholic acid

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Peritoneal membrane function | 6 months
  Changes in peritoneal membrane function (Δ D/Pcreatinine, ΔD/Purea) with peritoneal equilibrium test

SECONDARY OUTCOMES:
Residula renal function | 6 months
  Changes in estimated GFR
Epithelial to Mesenchymal Transition, EMT | 6 months
  Phenotypic changes of Mesothelial cells
Oxydative stress | 6 months
  Measurement of GSH/GSSG, 8-OHdG

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hee Kang, MD. PhD., Principal Investigator — Ewha Womans University Mokdong Hospital